CLINICAL TRIAL: NCT00321139
Title: An Assessment of Translesional Markers and Metabolomics
Brief Title: Assessment of Translesional Markers and Metabolomics
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Other Study IDs: 1189-2005
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Artery Disease
Keywords: biomarkers; oxidative stress; intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Blockages in the blood vessels of the heart are the main cause of chest pain, heart attacks, and sudden death. A cardiac catheterization, or injecting x-ray dye into the blood vessels of the heart and taking pictures, is currently the best way of assessing these blockages. This procedure, however, does not allow us to know what is happening inside the blockages. Some blockages have a higher risk of "rupturing" and completely blocking of the blood vessel while others are at low risk for doing this.

Blood levels of different substances produced by the body have been shown to be associated with a higher risk of having chest pain, a heart attack, or sudden death. There is also evidence from studies in animals and tissues taken from humans during surgery that some of these substances are made in the blockages themselves.

We would like to investigate whether a number of these substances are made in the blockages and released into the bloodstream. We will do this by taking one tablespoon samples of blood upstream and downstream of the blockages in the blood vessels of the heart. The samples will be obtained by using a very thin catheter, or plastic tubing, that is about 1/3 the size of the blood vessels of the heart. We will take samples from the tightest blockage found as well as another, less tight, blockage and compare the two. We will also sample blood from the tightest blockage after it is opened by doing an angioplasty. Finally, we will also take pictures of the blockages studied using a very small ultrasound camera inserted into the blood vessel. We will compare the levels of the substances measured with the features we see on the pictures.

We hope to learn if some or all of the substances measured can identify which blockages are more at risk for rupturing and causing heart attacks and sudden death.

All patients who are entered into this study will already be having an angioplasty done. The procedures needed for the study (sampling of blood and taking pictures with an ultrasound) are already often, though not always, used in patients undergoing an angioplasty.

DETAILED DESCRIPTION:
Introduction

Hypothesis

Coronary heart disease is the leading cause of death in the United States, accounting for > 500,000 lives each year. Atherosclerosis is the underlying mechanism for unstable angina, myocardial infarction, and sudden cardiac death. Luminal narrowing of the arteries caused by atherosclerotic plaque encroachment causes the chronic ischemic manifestations of coronary heart disease, whereas superimposition of thrombi over the plaques leads to acute coronary syndromes. To date, angiography has been the method of choice of detecting arterial lesions. However, this diagnostic technique, which approximately compares the degree of luminal stenosis of arteries relative to its' segments, does not provide insight into the disease state within the artery, and often fails to detect those lesions prone to thrombosis, often referred to as 'vulnerable plaque'. Multiple invasive and non-invasive methods have been employed in order to identify vulnerable plaque, usually by trying to image the plaque and its morphology, however none has gained widespread use.

Elevation of several biochemical markers in the bloodstream has been associated with adverse cardiovascular events. Inflammation has been identified as a significant component of the unstable atherosclerotic plaque. The inflammatory response seems to participate early in the development of atherosclerosis and involves multiple pathways3. Indeed, many markers of inflammation have now been shown to predict cardiovascular risk4-7 and recent studies have shown that key inflammatory markers are synthesized within atherosclerotic lesions8-10. Another process that appears to precede inflammation is oxidative stress. Increased cellular oxidative stress may be the process that initiates much of the subsequent inflammation and ultimately to development of the atherosclerotic process. Our preliminary data demonstrates that oxidative stress is increased in patients with acute coronary syndromes and after coronary stenting. The immune system is also activated in those with unstable atherosclerotic plaque with well documented changes in the T cells11-12.

An exciting new field of medicine is the application of systems approaches. One of these systems approaches is metabolomics. Metabolomics is based on the use of NMR (and other spectroscopic methods) and multivariate statistics for data analysis and interpretation. NMR spectroscopy is based on the behavior of atoms placed in a static external magnetic field. 1H-NMR spectroscopy allows the simultaneous detection and quantification of thousands of low-molecular-weight metabolites within a biologic fluid, resulting in the generation of an endogenous profile that may be altered in disease to provide a characteristic "fingerprint" of the disease process. It has been used clinically in the detection of ovarian cancer and coronary artery disease13, 14.

With this in mind, the difference in levels of oxidation and inflammatory markers, activated leucocytes, and the metabolomic profile across an atherosclerotic lesion, that is the translesional gradient, may be of clinical utility. An elevated translesional gradient of inflammatory and oxidative markers, leucocyte activation, as well as a change in the metabolomic profile, could be used to identify plaques prone to rupture. By implication, the ability to simply and reliably identify such plaques would have profound clinical consequences by either allowing placement of intracoronary stents in high-risk, but not yet flow-limiting lesions that if left untreated would rupture and lead to an acute coronary syndrome.

We hypothesize that:

1. the translesional gradients of (a) markers of oxidative stress, and (b) inflammation, and (c) activated leucocytes will be elevated across culprit lesions as opposed to non-culprit lesions in the same individuals; and
2. the translesional gradients of markers of oxidation, inflammation and leucocyte activation will differ in plaques with high-risk morphologic appearance compared to plaques with low-risk morphologic appearance, as assessed by intravascular ultrasound (IVUS); and
3. The metabolomic profile assessed by 1H-NMR spectroscopy will differentiate culprit and non-culprit lesions as well as plaques that have high-risk and low-risk morphologies.

Objectives

Aim 1: To determine and compare the translesional gradients of established markers of oxidative stress, inflammation, and leucocyte activation across culprit lesions vs non-culprit lesions in the same individuals.

Aim 2: To compare the translesion gradients of markers of oxidation, inflammation and leucocyte activation with plaque morphology as assessed by intravascular ultrasound (IVUS).

Aim 3: To determine if a systems approach using 1H-NMR-based metabolomics can be used to distinguish ruptured culprit and non-culprit lesions as well as plaques that have high-risk and low-risk morphologies.

Endpoints

1. A comparison of the markers of oxidation, inflammation, and leucocyte activation in the following:

   1. A comparison will be made between the translesional marker gradients (distal level - proximal level) of samples from the culprit lesion and non-culprit lesion.
   2. A comparison will be made between levels (distal level - proximal level) to the culprit lesion before and after angioplasty/stenting.
2. A comparison of the markers of oxidation, inflammation, and leucocyte activation with plaque morphologic indices as assessed by intravascular ultrasound.
3. A comparison of 1H-NMR metabolomic spectra from culprit and non-culprit lesions as well as plaques that have high-risk and low-risk plaque morphologies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from the ages of 21 and older
* Able to give informed consent
* Already scheduled to undergo diagnostic catheterization or percutaneous coronary intervention
* A culprit lesion (>60% diameter stenosis) in an artery that is at least 2.5 mm in diameter immediately proximal to the lesion.
* Presence of a second, non-culprit lesion, that is between 20 and 60% diameter stenosis in an artery that is at least 2.5 mm in diameter immediately proximal to the lesion.

Exclusion Criteria:

* ST-segment elevation myocardial infarction
* Thrombolysis in Myocardial Infarction (TIMI) grade 0 flow in the vessel containing the culprit lesion
* Autoimmune diseases, malignancy, or with active infections
* Taking immune-modulating therapies, eg prednisone
* Culprit lesion is in-stent restenosis
* Culprit lesion cannot be crossed with a wire and/or balloon
* Those enrolled in another research study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
A comparison of the markers of oxidation, inflammation, and leucocyte activation in the following:
A comparison will be made between the translesional marker gradients (distal level - proximal level) of samples from the culprit lesion and non-culprit lesion.
A comparison will be made between levels (distal level - proximal level) to the culprit lesion before and after angioplasty/stenting.
3. A

SECONDARY OUTCOMES:
A comparison of the markers of oxidation, inflammation, and leucocyte activation with plaque morphologic indices as assessed by intravascular ultrasound.
comparison of 1H-NMR metabolomic spectra from culprit and non-culprit lesions as well as plaques that have high-risk and low-risk plaque morphologies.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyad B Ghazzal, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States